CLINICAL TRIAL: NCT06266910
Title: Exploring the Effects of Autostereoscopic 3D Visual Training on Binocular Vision Function of Myopes Based on EEG and fNIRS
Brief Title: Effects of Autostereoscopic 3D Visual Training on Binocular Vision Function of Myopes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: South China University of Technology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023KYPJ320
Record Dates: First submitted 2024-02-01; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Myopia
Keywords: Myopia; Binocular visual function; Brain network; Neurovascular connectivity
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: By employing a single simulation technology for blinding, both the 2D group and the 3D group share identical training equipment and a consistent video background. The only distinction lies in the subtle variation in the configuration of training markers. It is difficult for participants to differentiate their respective groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three-dimensional (3D) viewing group (Experimental): Participants in this group watch a 10-minute training video displayed in 3D mode, twice a day (totaling 20 minutes), five days a week, for four consecutive weeks.
  Interventions: Other: Visual training video
- Two-dimensional (2D) viewing group (Placebo Comparator): Participants in this group watched a 10-minute training video displayed in 2D mode, twice a day (totaling 20 minutes), five days a week, for four consecutive weeks.
  Interventions: Other: Visual training video

INTERVENTIONS:
Other: Visual training video — The video, designed according to the principles of pencil pushups, features a dynamic standard "E" and is presented on an autostereoscopic 3D display equipment.

SUMMARY:
This study intends to conduct a relatively comprehensive binocular visual function examination and follow-up on two groups of myopic subjects, one receiving autostereoscopic 3D vision training and the other receiving 2D vision training as a control. The aim is to explore the impact of autostereoscopic 3D vision training on the accommodation and convergence functions of myopes. Additionally, synchronized EEG-fNIRS signals will be collected to investigate whether changes in binocular visual function are accompanied by corresponding alterations in brain function.

DETAILED DESCRIPTION:
The prevalence of myopia is increasing, posing a serious threat to our visual health. East Asia and Southeast Asia are high-prevalence areas for myopia, with over 80% of young people suffering from myopia. China has one of the highest rates of myopia globally. Preventing myopia occurrence and controlling its progression have become urgent public health issues.

Accommodative function may play an important role in the development of myopia. Studies indicate that factors such as hyperopic defocus caused by accommodation lag, prolonged near-plane fixation, and decreased accommodative flexibility may be associated with the occurrence and development of myopia. Convergence function works synergistically with accommodative function, and its impact on myopia is gradually gaining attention. Scientific and effective training methods to improve both accommodation and convergence functions might help slow down the progression of myopia.

Research by Huang et al. suggests that visual training based on autostereoscopic 3D display technology can improve accommodative lag and enhance accommodative flexibility. However, this study only explored the immediate effects of a single training session, and the long-term effects remain unknown. Furthermore, questions about how training induces changes in the convergence function, whether changes in accommodative function coincide with changes in the convergence function, etc., still need further investigation.

Therefore, this study intends to conduct a relatively comprehensive binocular visual function examination and follow-up on two groups of myopic subjects, one receiving autostereoscopic 3D vision training and the other receiving 2D vision training as a control. The aim is to explore the impact of autostereoscopic 3D vision training on the accommodation and convergence functions of myopes. Additionally, synchronized EEG-fNIRS signals will be collected to investigate whether changes in binocular visual function are accompanied by corresponding alterations in brain function.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 to 30 years
2. Refractive errors:

   spherical: -9.00 to -0.50 diopters (D), cylindrical: -2.50 to -0 D, and binocular difference within 2.0 D
3. Monocular best-corrected visual acuity ≥20/20
4. Normal stereoacuity
5. Participants capable of understanding the purpose of this study and providing informed consent
6. Participants capable of cooperating with relevant examinations.

Exclusion Criteria:

1. History of ophthalmic disease other than refractive error, such as strabismus, cataracts, glaucoma, retinal or optic nerve diseases
2. Use of any medications affecting accommodative function or wearing orthokeratology lenses in the past 1 month
3. History of ocular trauma or surgery
4. Suffering from systemic or mental illnesses.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Accommodative facility | 8 weeks after intervention
  Accommodative facility was tested using a lens flipper (+2.00D/-2.00 D lens combination) at baseline and 1 day, 1 week, 2 weeks, 4 weeks, and 8 weeks after intervention.
Vergence facility | 8 weeks after intervention
  Vergence facility was tested using a lens flipper (3△BI/12△BO lens combination) at baseline and 1 day, 1 week, 2 weeks, 4 weeks, and 8 weeks after intervention.

SECONDARY OUTCOMES:
Negative and positive fusional vergence | 8 weeks after intervention
  Negative and positive fusional vergence were measured by phoropter at baseline and 1 day, 1 week, 2 weeks, 4 weeks, and 8 weeks after intervention.
Accommodative response | 8 weeks after intervention
  Accommodative response was measured by the FCC method at baseline and 1 day, 1 week, 2 weeks, 4 weeks, and 8 weeks after intervention.
negative and positive relative accommodation | 8 weeks after intervention
  Negative and positive relative accommodation was measured by phoropter at baseline and 1 day, 1 week, 2 weeks, 4 weeks, and 8 weeks after intervention.
Near point of convergence | 8 weeks after intervention
  Near point of convergence was measured using push-up method at baseline and 1 day, 1 week, 2 weeks, 4 weeks, and 8 weeks after intervention.
Accommodation amplitude | 8 weeks after intervention
  Accommodative amplitude was measured by push-up method at baseline and 1 day, 1 week, 2 weeks, 4 weeks, and 8 weeks after intervention.
Electroencephalogram (EEG) node efficiency | 8 weeks after intervention
  Electroencephalogram was performed to track the electrical activity of the brain in real time at baseline and 1 day, 1 week, 2 weeks, 4 weeks, and 8 weeks after intervention. Node efficiency was calculated. Node efficiency is a metric that characterizes the efficiency of a single node in connecting with all other parts of the network. It reflects the centrality and importance of a node within the network.
Functional near-infrared spectroscopy (fNIRS) | 8 weeks after intervention
  Functional near-infrared spectroscopy (fNIRS) was conducted to capture spatial information on cerebral blood flow and oxygenation conditions at baseline, as well as 1 day, 1 week, 2 weeks, 4 weeks, and 8 weeks after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Opthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han J, Hong S, Lee S, Kim JK, Lee HK, Han SH. Changes in fusional vergence amplitudes after laser refractive surgery for moderate myopia. J Cataract Refract Surg. 2014 Oct;40(10):1670-5. doi: 10.1016/j.jcrs.2014.01.043. Epub 2014 Aug 20. PMID 25149555
- [Background] Tsujimoto K, Mizuno K, Nishida D, Tahara M, Yamada E, Shindo S, Watanabe Y, Kasuga S, Liu M. Correlation between changes in functional connectivity in the dorsal attention network and the after-effects induced by prism adaptation in healthy humans: A dataset of resting-state fMRI and pointing after prism adaptation. Data Brief. 2018 Dec 18;22:583-589. doi: 10.1016/j.dib.2018.12.053. eCollection 2019 Feb. PMID 30627613
- [Background] Wilf M, Serino A, Clarke S, Crottaz-Herbette S. Prism adaptation enhances decoupling between the default mode network and the attentional networks. Neuroimage. 2019 Oct 15;200:210-220. doi: 10.1016/j.neuroimage.2019.06.050. Epub 2019 Jun 22. PMID 31233909
- [Background] Ang M, Flanagan JL, Wong CW, Muller A, Davis A, Keys D, Resnikoff S, Jong M, Wong TY, Sankaridurg P. Review: Myopia control strategies recommendations from the 2018 WHO/IAPB/BHVI Meeting on Myopia. Br J Ophthalmol. 2020 Nov;104(11):1482-1487. doi: 10.1136/bjophthalmol-2019-315575. Epub 2020 Feb 26. PMID 32102791
- [Background] Huang Y, Li M, Shen Y, Liu F, Fang Y, Xu H, Zhou X. Study of the Immediate Effects of Autostereoscopic 3D Visual Training on the Accommodative Functions of Myopes. Invest Ophthalmol Vis Sci. 2022 Feb 1;63(2):9. doi: 10.1167/iovs.63.2.9. PMID 35113140
- [Background] Zhu Z, Chen Y, Tan Z, Xiong R, McGuinness MB, Muller A. Interventions recommended for myopia prevention and control among children and adolescents in China: a systematic review. Br J Ophthalmol. 2023 Feb;107(2):160-166. doi: 10.1136/bjophthalmol-2021-319306. Epub 2021 Nov 29. PMID 34844916